CLINICAL TRIAL: NCT02404142
Title: Curarisation and Intubation Conditions During Videolaryngoscopy With Glidescope Titanium
Acronym: GICAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHU de Reims (Other)
Collaborators: Verathon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI14034
Record Dates: First submitted 2015-03-17; First posted 2015-03-31 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Tracheal Intubation
Keywords: Trachel intubation; IDS score; Videoaryngoscopy; Glidescope® Titanium®; NMBA; Curare (Atracurium)
MeSH Terms: interventions — Curare; Atracurium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (saline isotonic solution) (Placebo Comparator): saline isotonic solution
  Interventions: Drug: saline isotonic solution
- Curar (Atracurium) group (Experimental): Curar (Atracurium)
  Interventions: Drug: Curare (Atracurium)

INTERVENTIONS:
Drug: Curare (Atracurium) — Curare (Atracurium) versus saline isotonic solution for tracheal intubation
  Arms: Curar (Atracurium) group
Drug: saline isotonic solution
  Arms: Control group (saline isotonic solution)

SUMMARY:
In this prospective, randomized study, the investigators assess the intubation conditions during videolaryngoscopy with Glidescope Titanium whether patients receive (curare (Atracurium) group) or no (control group) within elective surgery patients with no difficult intubation prediction

DETAILED DESCRIPTION:
In this prospective, randomized study, the investigators assess the intubation conditions during videolaryngoscopy with Glidescope Titanium whether patients receive (curare (Atracurium)group) or no (control group) within elective surgery patients with no difficult intubation prediction. The IDS score assessed by an anesthesiologist from the video-recording is the primary outcome. All general anesthesias are standardized using Target Control Infusion of propofol and sufentanil. The investigators also compare IDS scores as assessed by intubators, time for tracheal intubation, and laryngeal morbidity in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Elective Surgery Adult Patients
* no difficult intubation prediction

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-02-20; Primary Completion 2016-04-05 (Actual); Study Completion 2016-08-05 (Actual)

PRIMARY OUTCOMES:
IDS score video-assessed as described by Adnet et al. Measurement will be made by 2 experts anesthesiologists for centralized reading | Assessment will be done at the end of the inclusions period (9 months)
  Number of IDS scores <2 are compared

SECONDARY OUTCOMES:
IDS score assesed by the intubator anesthesiologist | 3 days post intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France